CLINICAL TRIAL: NCT03384264
Title: Changes in Phase Angle and Handgrip Strength Induced by Suspension Training in Older Women: A Randomized Controlled Trial
Brief Title: Effect of Suspension Training in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francesco Campa (Other)
Responsible Party: Sponsor-Investigator, Francesco Campa, Doctor, University of Bologna
Organization: University of Bologna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 28102016
Record Dates: First submitted 2017-12-19; First posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Effects of Suspension Training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TG (Experimental)
  Interventions: Other: Physical activity
- CG (No Intervention): the CG maintained their normal physical activity habits over the study

INTERVENTIONS:
Other: Physical activity — The suspension device was securely attached to a fixed beam. The suspension programme included an initial 10 min warm-up with very low-intensity joint mobility exercises. The central part of the program had a duration of 40 min and included six exercises in which the level of intensity was based on the inclination of the body. The exercises were performed in a split routine, alternating by segment to prevent joint overload. Finally, participants performed 10 minutes of stretching.
  Arms: TG

SUMMARY:
This study aimed to analyze the effects of a 12-week suspension exercise training programme on handgrip strength (HG) and anthropometric and bioelectrical impedance parameters in older adults.

ELIGIBILITY:
Inclusion Criteria:

non-hypertensive and not receiving hormonal replacement therapy,

Exclusion Criteria:

performing any regular physical exercise more than once a week over the 6 months preceding the beginning of the study

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Phase angle | 12 weeks
  Bioelectrical impedance parameter
Body composition | 12 weeks
  anthropometric measures
Handgrip strength | 12 weeks
  strength